CLINICAL TRIAL: NCT03132155
Title: A Phase 2 Study of AMG 337 in Subjects With Advanced or Metastatic Clear Cell Sarcoma That Contains the Ewing Sarcoma Breakpoint Region 1-activating Transcription Factor-1 (EWSR1-ATF1) Gene Fusion
Brief Title: QUILT-3.031: AMG 337 in Subjects With Advanced or Metastatic Clear Cell Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Prematurely terminated due to lack of therapeutic effect
Sponsor: NantPharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.031
Record Dates: First submitted 2017-04-20; First posted 2017-04-27 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Clear Cell Sarcoma
MeSH Terms: conditions — Sarcoma, Clear Cell | interventions — AMG 337

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMG 337 (Experimental): AMG 337 will be administered in patients with advanced or metastatic clear cell sarcoma
  Interventions: Drug: AMG 337

INTERVENTIONS:
Drug: AMG 337 — 6-{(1R)-1-[8-fluoro-6-(1-methyl-1H-pyrazol-4-yl)[1,2,4]triazolo[4,3-a]pyridin-3-yl]ethyl}-3-(2-methoxyethoxy)-1,6-naphthyridin-5(6H)-one•hydrate (1:1)

SUMMARY:
This is a phase 2 study that will assess the efficacy of AMG 337 in subjects with advanced or metastatic clear cell sarcoma that contains the EWSR1-ATF1 gene fusion.

DETAILED DESCRIPTION:
The phase 2 single arm study will assess efficacy of AMG 337 (based on confirmed ORR) in subjects with advanced or metastatic clear cell sarcoma that contains the EWSR1-ATF1 gene fusion, as determined by fluorescent in situ hybridization (FISH) or other diagnostic methods and confirmed by RNA sequencing (RNAseq).

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and provide a signed informed consent that fulfills the relevant Institutional Review Board (IRB) or Independent Ethics Committee (IEC) guidelines.
2. Able to attend required study visits and return for adequate follow-up, as required by this protocol.
3. Able to self-administer AMG 337 as a whole capsule by mouth every day.
4. Age ≥ 16 years.
5. Histologically confirmed, unresectable, locally advanced or metastatic tumors that contain the EWSR1-ATF1 gene fusion, as determined by fluorescent in situ hybridization (FISH) or other diagnostic methods and confirmed by RNA sequencing (RNAseq).
6. Have measurable disease evaluable in accordance with RECIST Version 1.1.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
8. Must have a recent Formalin-fixed paraffin-embedded (FFPE) tumor biopsy specimen that was obtained following the conclusion of the most recent anticancer treatment. If an historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period.
9. Must be willing to undergo a biopsy during the treatment period, if considered safe by the investigator.
10. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
11. Hematologic function, as follows:

    1. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L.
    2. Platelet count ≥ 50 × 109/L.
    3. Hemoglobin > 8 g/dL.
    4. Prothrombin time (PT) or partial thromboplastin time (PTT) < 1.5 × upper limit of normal (ULN), except for subjects on anticoagulation therapy for venous thromboembolism.
12. Renal function, as follows:

    a. Calculated creatinine clearance > 30 mL/min.
13. Hepatic function, as follows:

    1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 × ULN and total bilirubin < 1.5 × ULN.
    2. Alkaline phosphatase (ALP) < 2 × ULN (≤ 5 × ULN if bone or liver metastases are present)
14. Agreement to practice effective contraception (both male and female subjects, if the risk of conception exists).

Exclusion Criteria:

1. Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.
2. Inability to attend required study visits and return for adequate follow-up, as required for this protocol.
3. Known hypersensitivity to any component of the study medication(s).
4. Women who are nursing, pregnant, or planning to become pregnant during the duration of the study.
5. Current diagnosis or history of a second neoplasm, except the following:

   a. Adequately treated non-melanoma skin cancer, curatively treated in situ disease, or other solid tumors curatively treated with no evidence of disease for ≥ 2 years.
6. History of bleeding diathesis.
7. Uncontrolled hypertension (systolic > 160 mmHg and/or diastolic > 100 mmHg) or clinically significant cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months before study day 1; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication.
8. Baseline ECG Fridericia's formula QTcF > 470 ms.
9. Active infection requiring intravenous (IV) antibiotics within 2 weeks before study day 1.
10. Significant gastrointestinal disorder (eg, Crohn's disease, ulcerative colitis, extensive gastrointestinal resection) that in the opinion of the Investigator may influence drug absorption.
11. Positive result of screening test for human immunodeficiency virus (HIV).
12. Evidence of acute hepatitis B and C. Subjects with chronic hepatitis B or C are eligible if their condition is stable and, in the opinion of the investigator, would not pose a risk to subject safety.
13. Toxicities from prior anti-tumor therapy not resolved to CTCAE Version 4.03 grade 0 or 1.

    a. Grade 2 toxicities from prior anti-tumor therapy that are considered irreversible (defined as having been present or stable for > 4 weeks), such as stable grade 2 peripheral neuropathy or ifosfamide-related proteinuria, may be allowed if they are not otherwise described in the exclusion criteria.
14. Participation in this study or in an investigational study and/or procedure with any molecularly targeted agents reported to inhibit Mesenchymal epithelial transition factor (MET) within 14 days before study day 1.
15. Anti-tumor therapy, including chemotherapy, antibody therapy, retinoid therapy, or other investigational therapy within 14 days before study day 1.
16. Therapeutic or palliative radiation therapy within 14 days before study day 1.
17. Major surgery within 28 days before study day 1.
18. Any comorbidity that in the opinion of the investigator may increase the risk of toxicity.
19. Concurrent or prior use of a strong CYP3A4 inhibitor within 14 days before study day 1, including the following: ketoconazole, itraconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, and voriconazole.
20. Concurrent or prior ingestion of grapefruit or grapefruit products, or other foods known to inhibit CYP3A4 within 7 days before study day 1.
21. Concurrent or prior use of strong CYP3A4 inducers within 28 days before study day 1, including the following: phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, or the herbal supplement St. John's Wort.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-09-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Chan Soon-Shiong Institute for Medicine, El Segundo, California
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AMG 337: Subjects self-administered AMG 337 orally (PO) twice a day (BID, approximately every 12 hours) in a fasted state.
  Dose level 0: 150 mg BID (300 mg/day total) AMG 337 will be administered in patients with advanced or metastatic clear cell sarcoma
Period: Overall Study
Arm/Group | AMG 337
Started | 8
Completed | 0
Not Completed | 8
Not completed — Lack of Efficacy | 6
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- AMG 337: AMG 337 was administered in patients with advanced or metastatic clear cell sarcoma
  AMG 337: 6-{(1R)-1-[8-fluoro-6-(1-methyl-1H-pyrazol-4-yl)[1,2,4]triazolo[4,3-a]pyridin-3-yl]ethyl}-3-(2-methoxyethoxy)-1,6-naphthyridin-5(6H)-one•hydrate (1:1)
Arm/Group | AMG 337
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (13.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
SUBJECTS WITH ADVANCED OR METASTATIC CLEAR CELL SARCOMA THAT CONTAINS THE EWSR1-ATF1 GENE FUSION [Count of Participants; unit: Participants] | 8

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 337
Number analyzed (Participants) | 8
Participants
  Partial Response | 1
  Stable Disease | 1
  Progressive Disease | 5
  Imaging not available to evaluate | 1

2. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events (Safety And Tolerability)
Description: To evaluate the safety of AMG 337 based on grade 3 or 4 non-hematologic toxicity.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 337
Number analyzed (Participants) | 8
Participants
  Subjects with at Least 1 Grade 3 or 4 non-hematologic toxicity | 6
  Subjects without Grade 3 or 4 non-hematologic toxicity. | 2

ADVERSE EVENTS:
Time Frame: Non-serious AEs were followed for 30 days after the subject's last dose of study treatment, up to 13 months. Non-serious grade 3 or 4 AEs were followed until resolution or stabilization, up to 13 months. All SAEs that had not resolved upon discontinuation of the subject's participation in the study were followed until recovered, recovered with sequelae, not recovered (death due to other cause), death (due to the SAE), lost to follow-up. All-cause mortality approximately 3 years.
Arm/Group | AMG 337
All-Cause Mortality (participants affected / at risk) | 4/8
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 337 (N=8)
Abdominal pain (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 1
Diverticulitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 337 (N=8)
Dry skin (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Headache (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Abdominal pain (Nervous system disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Oedema (General disorders) | 2
Disease progression (General disorders) | 1
Facial pain (General disorders) | 1
Fatigue (General disorders) | 1
Influenza like illness (General disorders) | 1
Pyrexia (General disorders) | 1
Xerosis (General disorders) | 1
Anxiety (Psychiatric disorders) | 1
Dissociation (Psychiatric disorders) | 1
Nightmare (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Flushing (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Photophobia (Eye disorders) | 1
Diverticulitis (Infections and infestations) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to low enrollment. Only the safety data is provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/55/NCT03132155/Prot_SAP_001.pdf